CLINICAL TRIAL: NCT04099004
Title: Neural Correlates of Knee Sensorimotor Control in Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Greg Myer, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001773; 2017-5776 (Other: CCHMC Institutional Review Board)
Record Dates: First submitted 2019-04-11; First posted 2019-09-23 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Patellofemoral Pain Syndrome; Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neural Imaging (Other): Females with PFP attending a single study visit where neural imaging is acquired via MRI.
  Interventions: Other: Neural Imaging

INTERVENTIONS:
Other: Neural Imaging — During the acquisition of magnetic resonance (MR) images, the study participants will lie on the scanner table. For most portions of MR acquisition, the study participants will be instructed to lie still. For other parts of the acquisition, study participants will be asked to complete a combined knee and hip flexion/extension movement and a quadriceps contraction task in which they will be asked to 'squeeze' their quadriceps while keeping the rest of their body still. For the last 15 minutes of MR acquisition, the researcher will place one hand above the participants' knee and apply intermittent pressure to their quadriceps and medial aspect of the patella. Pain scales will be administered after every fMRI task to assess subjective perceptions of pain. Peripheral pulse oximetry and respiration waveforms will be collected for data analysis in order to minimize the potential confounding effect from the physiological changes.

SUMMARY:
This study aims to determine the neural correlates of knee motor control in young females with patellofemoral pain (PFP). Each participant will attend a single study visit which may last up to 3 hours.

DETAILED DESCRIPTION:
Patellofemoral pain (PFP) is one of the most common reported knee conditions in adolescents and young adults. PFP can affect nearly 30% of young adults and most frequently affect those who participate in athletic activities involving running, jumping, and cutting. Pain during movement also adversely influences patellofemoral joint loading as evidenced by increased frontal and transverse plane hip motion during activities of daily living. While the biomechanical and anatomical components contributing to knee pain have been well established, the underlying neural mechanisms are less understood. For adults with chronic pain (e.g., osteoarthritis), patients often exhibit greater 'pain network (e.g., anterior cingulate cortex, thalamus)' activation during sensory testing relative to healthy controls, possibly due to long term peripheral receptor activation resulting in hypersensitivity. Further, inducing pain (e.g., pressing on a thumbnail) results in similar neural activation of the pain network for those who have chronic pain symptoms.

While these studies have been imperative to the understanding of pain on neural functioning, they are limited to those specific populations (e.g., fibromyalgia, osteoarthritis) and do not adequately replicate the pain experienced during daily activities. Traditional approaches consisting of bracing and physical therapy focused on strengthening the knee extensors have been unsuccessful in reducing pain. Further, interventions consisting of exercise therapy have not been effective for all patients with PFP, and other pain-reduction techniques, such as direct electrical stimulation of the motor cortex, have failed to produce improved motor function or long-lasting pain relief. The researchers of this study hypothesize that this is due to the failure to appropriately challenge the full sensorimotor network involved in processing sensory and cognitive stimuli for motor control. To effectively treat pain and manage this condition, the neural correlates of pain and sensorimotor knee control in those with PFP is needed.

To appropriately assess the pain network for those with PFP, replicating knee and hip motion while neural function is measured is needed. The research team has successfully developed a combined knee and hip extension and flexion task that can be used safely with functional magnetic resonance imaging (fMRI). The researchers hypothesize that those with PFP will display depressed sensorimotor activity and increased pain network activity during the knee and hip flexion and extension task relative to previously collected data.

The study visit will consist of one magnetic resonance imaging (MRI) session using a GE SIGNA™ Premier 3.0 Tesla MR scanner. The MRI portion of the study visit will be completed in 75 minutes or less, and the entire visit will last up to 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with patellofemoral pain (PFP) or anterior knee pain by a medical professional
* Able to provide written consent

Exclusion Criteria:

* Any contraindications to MRI

Ages: 7 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Resting State Blood Oxygen Level Dependent (BOLD) Signal | Day 1 (during MRI session)
  Brain activity while the participant is lying still will be assessed as the BOLD signal obtained using fMRI.
Blood Oxygen Level Dependent (BOLD) Signal During Flexion/Extension Movement | Day 1 (during MRI session)
  Brain activity while participants complete a combined knee and hip flexion/extension movement will be assessed as the BOLD signal obtained using fMRI.
Blood Oxygen Level Dependent (BOLD) Signal During Quadriceps Contraction | Day 1 (during MRI session)
  Brain activity while participants complete a a quadriceps contraction task will be assessed as the BOLD signal obtained using fMRI. For the quadriceps contraction task, participants are asked to 'squeeze' their quadriceps while keeping the rest of their body still.
Blood Oxygen Level Dependent (BOLD) Signal During Pain Inducing Tasks | Day 1 (during MRI session)
  Brain activity while participants complete pain inducing tasks will be assessed as the BOLD signal obtained using fMRI. The pain inducing tasks involve the researcher placing one hand above the participants' knee and applying intermittent pressure to their quadriceps and medial aspect of the patella.

SECONDARY OUTCOMES:
Pain Scale Score | Day 1 (during MRI session)
  Participants reporting experiencing pain lasting longer than several days in the past two weeks complete a 4-item survey rating current, average, lowest and highest pain levels. Responses are given on a 5-point scale where 1 = no pain and 5 = worst pain possible. Total scores range from 4 to 20 and higher scores indicate greater pain.
Anterior Knee Pain Scale (AKPS) Score | Day 1 (during MRI session)
  Perceived movement dysfunction and disability related to knee pain is assessed using the Anterior Knee Pain (AKPS) scale. The AKPS has 13 items that are scored on scales of 0 to 5 or 0 to 10. Total scores range from 0 to 100 with 100 indicating the best knee function possible.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form Score | Day 1 (during MRI session)
  Perceived movement dysfunction and disability related to knee pain is assessed using the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form. The IKDC is a 10-item, patient-completed tool which contains sections on knee symptoms, knee function, and sports activities. Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Tampa Scale of Kinesiophobia (TSK) Score | Day 1 (during MRI session)
  Participant perceived movement dysfunction and disability related to knee pain is assessed using the Tampa Scale of Kinesiophobia (TSK). The TSK is a 17-item questionnaire assessing the fear of movement and re-injury. Responses are given on a 4-point Likert scale where 1 = strongly disagree and 4 = strongly agree. Total scores range from 14 to 68 where higher scores indicate greater concern of re-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Healthcare Sports Performance And Research Center (SPARC), Flowery Branch, Georgia
  - Cincinanti Childrens Hospital Medical Center (CCHMC), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT04099004/Prot_000.pdf